CLINICAL TRIAL: NCT02858622
Title: Unilateral Dual Transversus Abdominis Plane Block in Pediatric Renal Transplant: A Randomized Control Study
Brief Title: Dual Transversus Abdominis Plane Block in Pediatric Renal Transplant: Effect on Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Mohamed Abd el moneim Soaida, MD, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SMS2016-1
Record Dates: First submitted 2016-04-05; First posted 2016-08-08 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Renal Failure
Keywords: pediatric; renal transplant; pain; dual TAB
MeSH Terms: conditions — Renal Insufficiency; Pain | interventions — Bupivacaine; Meperidine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dual TAB group (Active Comparator): 22 patients will receive unilateral dual transversus abdominis plane (TAB) block USING bupivacaine 0.25% at a dose of 2 mg/kg
  Interventions: Drug: bupivacaine; Drug: Pethidine; Drug: perfalgan; Drug: fentanyl
- control group (Sham Comparator): 22 patients who will not receive dual TAB block
  Interventions: Drug: Pethidine; Drug: perfalgan; Drug: fentanyl

INTERVENTIONS:
Drug: bupivacaine — bupivacaine 0.25% at a dose 2 mg/kg in the transversus abdominis plane
  Arms: dual TAB group
Drug: Pethidine — pethidine intravenous at a dose 1mg/kg when pain score more than 5 postoperative rescue analgesia
Drug: perfalgan — intravenous paracetamol
Drug: fentanyl

SUMMARY:
Alleviating pain in children undergoing renal transplant is extremely challenging. Large incisions as those of renal transplant (Gibson's incision) require special techniques of pain control that don't affect hemodynamics or renal function. Since the transplant incision doesn't cross midline; a dual-TAP block is thought to be effective in providing pain control in such procedure as it will anesthetize the dermatomes T6-T12, the muscles of the anterior abdominal wall together with the underlying parietal peritoneum.

ELIGIBILITY:
Inclusion Criteria:

* 3-16 years
* end stage renal disease
* no known allergy to bupivacaine
* both sexes

Exclusion Criteria:

* known allergy to bupivacaine

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2016-12; Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
total dose of rescue analgesia | from the time of transfer of the patient to the intensive care unit at one hour intervals for 24 hours
  pethidine given as rescue analgesia postoperative.

SECONDARY OUTCOMES:
pain scoring system (objective behavioural pain score) | from the time of transfer to the nephrology ICU, every hour for the first 24 hours postoperative
Intraoperative blood pressure | from the induction of anesthesia till end of surgery at half an hour intervals average duration is 4 hours
  measure systolic and diastolic blood pressure
postoperative blood pressure | from the time of transfer of the patient to the intensive care unit at one hour intervals for 24 hours
  record systolic and diastolic blood pressure every hour for the first 24 hours postoperative
postoperative heart rate | from the time of transfer of the patient to the intensive care unit at one hour intervals for 24 hours
intraoperative heart rate | from the induction of anesthesia till end of surgery at half an hour intervals average duration is 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M Soaida, M.D., Principal Investigator — Cairo University
Locations (1):
- Faculty of medicine, Cairo University, Cairo, Egypt